CLINICAL TRIAL: NCT03688867
Title: Prehabilitation in Pancreatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4218
Record Dates: First submitted 2018-09-04; First posted 2018-09-28 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Resection; Preoperative Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At-home prehabilitation regimen (Experimental): 1. Grip strength: Squeeze a stress ball in your hand, holding it squeezed for 5 seconds. Perform this at least thirty times with each hand over the course of a day.
  2. Lower body strength: Perform at least one hundred chair sit-stands in a day.
  3. Endurance: Walking at least 7,500 steps in a day.
  Interventions: Behavioral: Prehabilitation regimen

INTERVENTIONS:
Behavioral: Prehabilitation regimen — The intervention targets individual behavior, specifically a patient's proclivity to exercise prior to pancreatic resection. The prehabilitation program is tailored to the three most commonly used objective frailty metrics currently available and will be implemented during the initial consultation visit in the surgery outpatient clinic, where patients will undergo baseline testing and then provided with a fitness tracker and stress ball.
  Additionally, they will be provided with an activity log to keep track of their daily activity. Shown below is the activity log.

SUMMARY:
The purpose of this study is to use functional studies to study the effectiveness of prehabilitation prior to surgery. The investigators know that stronger patients have better outcomes after surgery compared to weaker patients. This study will help the study team determine if prehabilitation can make patients stronger prior to surgery. It is hoped by learning more about frailty and prehabilitation strategies may be developed to minimize or prevent complications in the future. Participants are being asked to participate in this study because they are going to have a pancreatic procedure.

DETAILED DESCRIPTION:
This study aims to determine if a prehabilitation program can improve three objective frailty metrics and to describe the level of physical activity of pancreatectomy patients prior to their planned resection. Patients undergoing pancreatectomy will undergo routine preoperative work up: Staging PET/CT Chest/Abdomen/Pelvis, and biochemical work up (CBC, CMP, CA 19-9, prealbumin/albumin).

During the initial consultation, the patients' resting vitals (including weight) will be recorded. They will then perform the grip strength, 30s CST, and 6MWT to establish their baseline frailty metrics. Available baseline laboratory values (CBC, CMP including albumin), will also be recorded. Research personnel will then provide them with a fitness tracker, stress ball, and prehabilitation routine to follow at home until the day of surgery. They will also be asked to keep a physical log of their completed physical activities.

The patients will then complete the prehabilitation program during the time between the initial consultation and date of surgery, which typically occurs 3-4 weeks after the initial consultation date.

On the day of surgery, patients will turn in their physical log and their fitness tracker. Data from the fitness tracker will be downloaded onto a Cleveland Clinic encrypted computer. A set of resting vitals will be recorded (again including weight) and the patients will then be asked to perform the three-frailty metrics (grip strength, 30s CST, and 6MWT). After this, the patients will not require any additional testing.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing pancreatic resection over a six-month enrollment

Exclusion Criteria:

* unable to sign a consent
* require a translator in order to sign the consent
* Non-pancreatic resection candidates

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Change in grip strength | 4 weeks
  Participant's grip strength will be measured before and after intervention with a Jamar Dynamometer as follows:
  1. Hold both arms at 90-degree angles with the arms held close to the body
  2. Perform isometric contraction for 5 seconds and measure the pressure generated from this
  3. Both handgrips will be measured three times each and averaged. The greater of the two averages will be recorded
Change in number of chair stands in 30 seconds (chair stand test) | 4 weeks
  The change in the number of times the participant can fully stand up from a seated position in 30 seconds will be measured as follows:
  Participant will
  1. Sit in the middle of the chair
  2. Place their hands on the opposite shoulder crossed at the wrists
  3. Keep their feet flat on the floor
  4. Keep their back straight and keep their arms against your chest
  5. On "Go," rise to a full standing position and then sit back down again
  6. Repeat this for 30 seconds
  7. If the participant must use his/her arms to stand, stop the test. A score of "0" will be recorded for the number and score. The number of times the patient comes to a full standing position in 30 seconds will be counted. If the patient is over halfway to a standing position when 30 seconds have elapsed, it will count as a stand. Number of times the patient stands in 30 seconds will be recorded.
Change in vitals and distance walked via 6-minute walk test | 4 weeks
  The change in the participant's 6-minute walk test metrics (vitals and distance walked)
  1. Participant's baseline vitals will be recorded, including pulse oximetry prior to walking
  2. Participant will walk as far as possible in 6 minutes at a comfortable pace, but not at a run or jog.
  3. If they become short of breath or tired, they may slow down, stop, or rest as necessary. Participant may lean against the wall while resting, but will resume walking as soon as they are able.
  4. Participant will walk down to the end of the hall, turn around and walk back. They will repeat this until the six minutes have expired.
  5. If the participant is unable to complete the full six-minute walk, then the time and distance walked will be recorded as well as the reason for stopping early.
  Vitals will be recorded immediately after walking

SECONDARY OUTCOMES:
Number of grip exercises | 4 weeks
  Participants will complete and record number of stress ball squeezes (Squeezing stress ball in hand and holding it squeezed for 5 seconds) during the prehabilitation period
  Number of times squeezed with right hand and number of times squeezed with left hand will be recorded.
Number of chair sit stands performed | 4 weeks
  Measures lower body strength: Participants will measure the number of chair sit stands they perform in a day during the prehabilitation period.
Number of steps walked | 4 weeks
  Participants will track the number of steps they walk per day during the prehabilitation period via the provided fitness activity tracker (Garmin Vivofit 4).
Heart rate | 4 weeks
  Participants will track their heart rate during the prehabilitation period via the provided fitness activity tracker (Garmin Vivofit 4).
Energy expenditure | 4 weeks
  Participant's energy expenditure will be tracked via the data from the supplied fitness tracker (Garmin Vivofit 4).
Weight change from the baseline | 4 weeks
  Participant's weight change from the baseline initial consultation to the day of operation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Walsh, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States